CLINICAL TRIAL: NCT05628168
Title: Effect of Neurodynamic Mobilization Techniques in Patients With Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Ahmed Magdy Alshimy, Lecturer of Physical Therapy at department of Neurology, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003496
Record Dates: First submitted 2022-11-13; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Diabetic Neuropathies
Keywords: Neurodynamic technique; Sensory nerve conduction study; Motor nerve conduction study; Functional outcome; Diabetic polyneuropathy.
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The NMG received three sessions/week for 4 weeks with each session lasting for 30 min including slider and tension neurodynamic techniques.
  Interventions: Other: Neurodynamic Mobilization Techniques; Other: Selected Physical Therapy Program
- Group B (Active Comparator): The participants only received a selected therapy program similar to the NMG with no change in duration.
  Interventions: Other: Selected Physical Therapy Program

INTERVENTIONS:
Other: Neurodynamic Mobilization Techniques — The slider neurodynamic technique for the median nerve is conducted.Tensioner neurodynamic technique for the tibial nerve is conducted.
  Arms: Group A
Other: Selected Physical Therapy Program — The participants only received a selected therapy program similar to the NMG with no change in duration.

SUMMARY:
Neurodynamic mobilization Techniques and Selected Physical program used as a treatment for diabetic neuropathy patients and assessed by nerve condition study and function outcome.

DETAILED DESCRIPTION:
Neurodynamic mobilization Techniques and Selected Physical program used as a treatment for diabetic neuropathy patients and assessed by nerve condition study and function outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2DM for ≥10 years determined by electrophysiological measurements were enrolled.
* The participants regularly took their diabetes medications during the assessment and treatment period.

Exclusion Criteria:

* Uncontrolled T2DM and diagnosed with T2DM for < 10 years.
* Patients with neural, muscular, and skeletal system deformities; radiculopathy; and psychiatric disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Effect of Neurodynamic Mobilization Techniques in Patients With Diabetic Neuropathy | 5-6 months
  This study aimed to investigate neurodynamic mobilization effect on sensory and motor nerve conduction study, pain, and functional activity in patients with type 2 diabetic neuropathy and will be assessed through Katz index and NIHON KODEN EMG device.

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No